CLINICAL TRIAL: NCT03216720
Title: The Impact of Miniaturized Extracorporeal Circulation on Thrombin Generation and Postoperative Blood Loss
Brief Title: Miniaturized Extracorporeal Circulation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Responsible Party: Principal Investigator, Ivy susanne Modrau, MD, Consultant Cardiac Surgeon, Associate Professor, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-16-02-188-17
Record Dates: First submitted 2017-07-08; First posted 2017-07-13 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery bypass grafting; Miniaturized extracorporeal circulation; Thrombin generation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CABG with miniaturized ECC (Active Comparator): Elective (CABG) with conventional miniaturized extracorporeal circulation (miECC)
  Interventions: Procedure: CABG; Procedure: Miniaturized extracorporeal circulation
- CABG with conventional ECC (Active Comparator): Elective CABG with conventional extracorporeal circulation (cECC)
  Interventions: Procedure: CABG; Procedure: Conventional extracorporeal circulation

INTERVENTIONS:
Procedure: CABG — * Cannulation: 24-F arterial cannula, 29/29 F dual-stage venous cannula, and aortic root vent-/cardioplegia cannula
  * Grafting: pedicled left internal mammary artery, and no-touch
  * saphenous vein graft Heparin and protamine doses assessed by HMS Plus® Hemostasis Management System
  * Target activated coagulation time of >400 seconds
Procedure: Miniaturized extracorporeal circulation — * Centrifugal pump to reduce mechanical stress
  * Circuit coated with biosurface to increase haemocompatibilty.
  * Ante- and retrograde autologous priming and low-volume cardioplegia solution (intermittend cold modified Calafiore) to minimize haemodilution
  * Collapsible soft-shell reservoir for blood volume management
  * Cell-saving device
  * Venous air removing device and electric clamp system to air embolism
  Arms: CABG with miniaturized ECC
Procedure: Conventional extracorporeal circulation — * Roller pump
  * Circuit uncoated
  * Hard-shell venous reservoir
  * Intermittend cold blood Harefield cardioplegia
  Arms: CABG with conventional ECC

SUMMARY:
Rationale:

Contemporary coronary artery bypass grafting (CABG) continues to be associated with a significant risk of postoperative bleeding. Utilization of miniaturized extracorporeal circulation (miECC) significantly reduces the risk of postoperative bleeding but the underlying mechanisms are poorly understood.

Primary Objective:

To assess the impact of miECC compared to conventional extracorporeal circulation (cECC) on thrombin generation as indicator of the overall haemostatic capacity after CABG.

Secondary Objectives To evaluate the impact of miECC versus cECC on blood loss and transfusion requirement, coagulation and fbrinolysis, inflammatory response, haemodilution and haemolysis, endorgan protection, seasibility and safety

Study design:

Single-center, double-blind, parallel-group randomized controlled trial

Study population:

60 Patients undergoing non-emergent primary isolated CABG with ECC randomized 1:1 to receive either miECC or cECC

DETAILED DESCRIPTION:
Blood samples will be obtained at the following time points:

* T0; preoperative after induction of anaesthesia (after insertion of central venous line)
* T1; after weaning of the ECC prior to protaminization
* T2; 10 minutes after full protaminization
* T3; six hours after the end of the ECC
* T4; 1. postoperative day (16-20 hours following end of surgery)

ELIGIBILITY:
Inclusion Criteria:

* Non-emergent CABG with ECC
* Current use of low-dose acetylsalicylic acid
* Agreement of eligibility by the multidisciplinary heart team

Exclusion Criteria:

* Inability to give informed consent
* Emergent treatment required (< 24 hours)
* Concomitant cardiac surgery
* Previous cardiac surgery
* Severely reduced kidney function (eGFR < 30ml/min/1.73m2 or on dialysis)
* Severely reduced ejection fraction (EF < 45%)
* Diagnosis of bleeding disorders
* Non-aspirin antiplatelet drugs stopped < 5 days preoperatively (Clopidogrel, Prasugrel, Ticagrelor, Ticlopidine)
* Current use of systemic glucocorticoid therapy
* Current use of vitamin K antagonists or new oral non-vitamin K anticoagulants
* Platelet count > 450 or <100 x 109/l prior to surgery
* Pregnant women or women of child bearing potential without negative pregnancy test
* Active participant in any other intervention trial

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Postoperative thrombin generation | up to 6 hours after CABG
  Thrombin generation as a measure of the ability to generate thrombin in platelet poor plasma. Derived from the thrombogram

SECONDARY OUTCOMES:
Postoperative blood loss | up to 24 hours after CABG
  Total output of mediastinal and pleural chest tubes
Postoperative transfusion requirement | up to 30 days after CABG
  Transfusion of red blood cells, fresh frozen plasma, platelets
Fibrinolysis (Clot lysis, Fibrin D-dimer) | up to 24 hours after CABG
  Clot lysis measured by dynamic turbidimetry
Coagulation tests | up to 24 hours after CABG
  * Platelet Count
  * aPTT
  * INR
  * Antithrombin
  * Fibrinogen
  * Prothrombin fragment 1+2
Inflammatory response | up to 24 hours after CABG
  * TNF-α
  * Interleukin panel
  * CRP white blood count
Haemodilution (Nadir intraoperative haematocrit) | up to 24 hours after CABG
  Measured in arterial blood samples
Haemolysis (LDH) | up to 24 hours postoperative
  Measured in lithium heparin plasma
Postoperative CK-MB for myocardial injury | up to 24 hours after CABG
  Measured in lithium heparin plasma
-Intraoperative blood lactate for inadequate tissue perfusion | up to 24 hours after CABG
  Measured in arterial blood samples
Postoperative creatinine clearance for renal injury | up to 30 days after CABG
  Creatinine measured in lithium heparin plasma. eGFR calculated according to the CKD EPI Equation for Estimating GFR Expressed for Specified Race, Sex and Serum Creatinine (µmol/L)
-Perioperative myocardial infarction | 48 hours after CABG
  defined according to the new definition of clinically relevant MI of the Society for Cardiovascular Angiography and Interventions
-In-hospital neurological events (TCI/stroke) | up to 30 days after CABG
  verified by CT or MRI
-Postoperative requirement of renal replacement therapy | up to 30 days after CABG
  Continuous or intermittend renal replacement therapy
-Postoperative re-exploration for bleeding | up to 30 days after CABG
  Re-exploration due to excessive bleeding or haemodynamic instability
-Repeat revascularization | up to 30 days after CABG
  Defined as unplanned repeat PCI or CABG
-Length of ICU stay | up to 30 days after CABG
  Days of stay on ICU
-Duration of inotropic support | up to 30 days after CABG
  Hours of pharmacological or mechanical circulatory support
-Incidence of atrial fibrillation | up to 30 days after CABG
  Documented by telemetry or ECG
-Incidence of infection (requiring antibiotic therapy, wound revision for graft leg infection, superficial or deep sternal wound infection) | up to 30 days after CABG
  * Deep sternal wound infection
  * Wound revision for leg harvest surgical site infection
  * Requirement of antibiotic therapy
-Feasibility of miECC as measured by conversion to cECC and intraoperative complications | 24 hours
  Serious adverse device events (air lock, dissection, bleeding that exceeds the capacity of the cell saver, air emboli, stop of the circuit, conversion to cECC)
  - technical aspects (postoperative fluid gain (ml), venous drainage, visibility due to blood in the operative field, ability to maintain SvO2 >65%)
-30-day MACCE | up to 30 days after CABG
  * Death
  * MI
  * cerebrovascular accident
  * repeat revascularization
Acute kidney injury | up to 7 days after intervention
  Association of AKI with Neutrophil gelatinase associated lipocalin (NGAL) and renal risistive index (RRI)

CONTACTS AND LOCATIONS:
Overall Officials: Ivy Susanne Modrau, MD, Principal Investigator — Dep. of Cardiothoracic Surgery, Aarhus University Hospital Skejby
Locations (1):
- Dep. of Cardiothoracic Surgery, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halle DR, Benhassen LL, Soberg KL, Nielsen PF, Kimose HH, Bauer A, Hasenkam JM, Modrau IS. Impact of minimal invasive extracorporeal circulation on systemic inflammatory response - a randomized trial. J Cardiothorac Surg. 2024 Jul 3;19(1):418. doi: 10.1186/s13019-024-02903-8. PMID 38961388
- [Derived] Modrau IS, Halle DR, Nielsen PH, Kimose HH, Greisen JR, Kremke M, Hvas AM. Impact of minimally invasive extracorporeal circulation on coagulation-a randomized trial. Eur J Cardiothorac Surg. 2020 Jun 1;57(6):1145-1153. doi: 10.1093/ejcts/ezaa010. PMID 32011717

DOCUMENTS (1):
  • Study Protocol (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT03216720/Prot_000.pdf